CLINICAL TRIAL: NCT02003638
Title: A 12-WEEK STUDY EVALUATING THE EFFECTS OF NIACIN ON VASCULAR HEALTH ASSESSED BY FLUORODEOXYGLUCOSE-PET/CT AND CIRCULATING ENDOTHELIAL PROGENITOR CELLS AND MICROPARTICLES
Brief Title: Assessment Of Vascular Health After Niacin Therapy (AVANT)
Acronym: AVANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Emil deGoma, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 812962
Record Dates: First submitted 2013-11-18; First posted 2013-12-06 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease; Carotid Artery Disease; Peripheral Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Carotid Artery Diseases; Peripheral Arterial Disease | interventions — Niacin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niacin (Experimental): Niacin titrated up to 6 grams taken orally every day for 12 weeks
  Interventions: Drug: Niacin
- Placebo (Placebo Comparator): Placebo taken orally every day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niacin — Niacin titrated to 6000 mg daily
  Other Names: Niaspan; Niacor
  Arms: Niacin
Drug: Placebo — Placebo provided in the same pill quantity as niacin arm
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study is looking to see if niacin will lessen atherosclerotic plaque inflammation and favorably affect circulating levels of endothelial progenitor cells and microparticles in people with atherosclerotic disease on chronic statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men age 55 years and above with coronary artery disease or women age 65 years and above with coronary artery disease OR Men age 45 years and above with both coronary artery disease and carotid or lower extremity peripheral artery disease or women age 55 years and above with both coronary artery disease and carotid or lower extremity peripheral artery disease.
* Subjects must be on statin monotherapy, defined as a stable statin dose for at least 12 weeks, with no anticipated need for further titration during the study period

Exclusion Criteria:

* Anxiety or claustrophobia prohibiting imaging
* History of allergy to intravenous contrast, iodine, or shellfish
* Renal insufficiency
* History of allergy or severe intolerance to niacin
* History of diabetes mellitus or elevated fasting glucose
* Moderate to severe gout
* Peptic ulcer disease
* Acute coronary syndrome, transient ischemic attack or cerebrovascular accident, or acute limb ischemia in the preceding 12 months
* Heart failure or unstable angina pectoris
* Use of daily non-statin lipid-altering therapy prior to the initiation of study medication

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil deGoma, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niacin | Placebo
Started | 6 | 3
Completed | 5 (1 withdrew after developing bacterial pharyngitis. Not considered treatment-emergent.) | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin | Placebo | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Full Range); unit: years] | 63 [56 to 67] | 66 [64 to 69] | 64 [56 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 3 | 8
Body-mass index [Mean (Full Range); unit: kg/m^2] | 28.9 [23.7 to 33.1] | 32 [25.6 to 33.4] | 30.0 [23.7 to 33.4]
Coronary artery disease [Number; unit: participants] | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Arterial Fluorodeoxyglucose (FDG) Uptake Assessed by FDG-PET/CT
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Target to Background Ratio (TBR)
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 5 | 3
Target to Background Ratio (TBR) | -0.02 (.14) | -0.05 (.12)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Niacin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 3/5 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin (N=5) | Placebo (N=3)
Abdominal pain (General disorders) | 1 (1) | 0 (0) — At week 11, hospitalized for abdominal discomfort, nausea, chest pain. Vital signs, serial ECG, cardiac enzymes, chest radiography, and hemoglobin were normal. His symptoms resolved spontaneously within 24 hours without cessation of study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niacin (N=5) | Placebo (N=3)
Rocky Mountain Spotted Fever (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Asymptomatic. Incidental finding of chronic pulmonary emboli on baseline CT

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No